CLINICAL TRIAL: NCT03499496
Title: Prevalence of Atherosclerotic Carotid and/or Femoral Plaques in Patients Without Known Cardiovascular Disease and at Low-risk for Major Cardiovascular Events (AGLA/GLSA Score) Visiting a Private Primary Healthcare Practice in Switzerland
Brief Title: Screening for Atherotic Plaques by Ultrasound for Assessing Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: Cabinet de Medecine Interne Générale Demetrio Pitarch (Other)
Responsible Party: Sponsor
Other Study IDs: DPitarch
Record Dates: First submitted 2018-03-22; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Atherosclerosis of Artery
Keywords: plaques detection by ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound guided detection of atherosclerotic plaques — screening by ultrasound of atherosclerotic plaques

SUMMARY:
Cardiovascular disease is a common diagnosed and treated condition in private practices of primary health care. There is growing evidence that atherosclerotic plaques as predictors for stroke and heart attack are more prevalent than expected based on the clinical score in people with low risk for stroke and heart attack .

Diagnosing atherosclerotic plaques can help to decide if a lipid lowering therapy should be prescribed even if the clinical risk score is low or on the other hand if they can be observed even in high lipid levels.

DETAILED DESCRIPTION:
Both common and proximal internal carotid arteries and both common femoral arteries (including bifurcations) were screened by ultrasound in patients who came for a check-up to a primary care practice with no known cardiovascular disease and low risk for stroke and heart attack according to the AGLA/GSLA risk score which is mostly used in Switzerland.

All patients agreed and gave written informed consent to be included in this study. Presence of plaques was defined as a focal carotid intima-media thickness >0.5 cm on ultrasound. Screening was performed by a medical doctor (DP) certified for the procedure using the following ultrasound system: Toshiba Nemio XG, probe 7.5 MhZ.

ELIGIBILITY:
Inclusion Criteria:

* low cardiovascular risk assessed by the AGLA/GSLA-score

Exclusion Criteria:

* cardiovascular disease

Ages: 41 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The carotid and femoral arteries of 22 asymptomatic patients (9 females,13 males) aged between 41-72 having a low cardiovascular risk score based on blood pressure, nicotine abuse history, cardiac family history, blood analysis in fasting state for diabetes, lipid status including total cholesterol HDL-cholesterol, triglycerides and calculated LDL-cholesterol were screened by ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-09-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of plaques in cardiovascular low risk population | 1 year
  Number of participants with the presence of carotid and/or femoral atherosclerotic plaques diagnosed via ultrasound (defined as a focal intima-media thickness >0.5 cm on ultrasound).

CONTACTS AND LOCATIONS:
Overall Officials: Demetrio A Pitarch, MD, Principal Investigator — Cabinet de medecine generale

IPD SHARING:
Plan to Share IPD: No